CLINICAL TRIAL: NCT00005792
Title: A Study of Intensive-Dose Melphalan, Topotecan, and VP-16 Phosphate (MTV) Followed by Autologous Stem Cell Rescue in Patients With Multiple Myeloma
Brief Title: Combination Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: SmithKline Beecham (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-11752; MCC-11752 (Other: Moffitt Cancer Center); IRB-4983 (Other: University of South Florida); NCI-G00-1749 (Other: National Cancer Institute)
Record Dates: First submitted 2000-06-02; First posted 2004-02-02 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma; Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — etoposide phosphate; Topotecan; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MTV (Experimental): Melphalan Topotecan Etoposide VP-16 Phosphate autologous stem cell transplant
  Interventions: Drug: etoposide phosphate; Drug: melphalan; Drug: topotecan; Procedure: Autologous Stem Cell Rescue

INTERVENTIONS:
Drug: etoposide phosphate — Etoposide phosphate 1363 mg/m^2/day IV over 4 hours (total dose 2726 mg/m^2, or 2400 mg/m^2 etoposide equivalents), beginning 24 hours after the completion of the last infusion of topotecan Days -4, -3
  Other Names: Topotecan
Drug: melphalan — Melphalan 50 mg/m^2/day IV over 30 minutes (total dose 150 mg/m^2), followed immediately by topotecan. Days -7, -6, -5
  Other Names: Alkeran(R)
Drug: topotecan — Topotecan 3.3 mg/m^2/day (starting total dose = 10 mg/m^2 for level 2) IV over 30 minutes. No topotecan will be administered on the first dose level Days -7, -6, -5
Procedure: Autologous Stem Cell Rescue — reinfusion of stem cells, Day 0
  Other Names: Autologous stem cell transplant

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy plus peripheral stem cell transplantation in treating patients who have multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity and potential efficacy of intensive high dose chemotherapy consisting of melphalan, topotecan, and etoposide phosphate followed by autologous stem cell transplantation in patients with stage II or III multiple myeloma or stage I with evidence of progressive disease. II. Determine the maximum tolerated dose of topotecan in combination with melphalan and etoposide phosphate in this patient population. III. Determine response rates and time to treatment failure in these patients when treated with this regimen. IV. Determine the pharmacokinetic profiles of these drugs and investigate the pharmacodynamic relationships with respect to the efficacy and toxicity of this regimen in these patients. V. Determine whether the sequencing of this chemotherapy regimen is appropriate and optimal in these patients.

OUTLINE: This is a dose escalation study of topotecan. Patients are primed with cyclophosphamide IV over 2 hours for 2 days. Peripheral blood stem cells (PBSC) are collected. Approximately 4 weeks after PBSC collection, patients receive melphalan IV over 30 minutes and topotecan IV over 30 minutes on days -7 to -5. Etoposide phosphate IV is administered over 4 hours on days -4 and -3. PBSC are reinfused on day 0. Cohorts of 4-12 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 6 of 12 patients experience dose limiting toxicities. Patients are followed 2-3 times a week for approximately 1 month, then at 3, 6, and 12 months.

PROJECTED ACCRUAL: A total of 34-60 patients will be accrued for this study within 24-36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed multiple myeloma Newly diagnosed, drug sensitive (i.e., greater than 50% response to standard chemotherapy), and poor prognostic indicators (e.g., Salmon-Durie stage III, serum beta-2-microglobulin greater than 3.0 ug/L, high proliferative fraction, or hypodiploidy) OR Relapsed after a response to standard chemotherapy OR Primary refractory disease No active leptomeningeal involvement History of prior CSF tumor involvement without symptoms or signs allowed provided CSF is now free of disease on lumbar puncture and MRI of brain shows no tumor involvement No severe symptomatic CNS disease of any etiology

PATIENT CHARACTERISTICS: Age: 15 to 69 Performance status: ECOG 0-1 ECOG 3-4 secondary to bone pain or a potentially reversible disease related problem eligible at investigator's discretion Life expectancy: At least 12 weeks Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT/SGPT no greater than 2.5 times upper limit of normal No history of severe hepatic dysfunction Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine at least 40 mL/min No hemodialysis or peritoneal dialysis Cardiovascular: No evidence of severe cardiac dysfunction Ejection fraction at least 50% by MUGA scan No major heart disease Essential hypertension controlled with medications allowed Pulmonary: DLCO at least 50% of normal No symptomatic obstructive or restrictive pulmonary disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No psychosocial disorder that would preclude study compliance No active infections No uncontrolled insulin dependent diabetes mellitus No uncompensated major thyroid or adrenal dysfunction No other prior malignancy except for nonmelanoma skin cancer HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior total dose of doxorubicin or daunorubicin greater than 450 mg/m2 No prior topotecan or any other topoisomerase I inhibitor, etoposide, etoposide phosphate, or teniposide Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No concurrent nitroglycerin preparations for angina pectoris No concurrent antiarrhythmic drugs for major ventricular dysrhythmias

Ages: 15 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 1998-06-02 (Actual); Primary Completion 2006-07-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of mucositis | 5 years
  To determine the incidence and duration of CTCAE v3, grade 3 or 4 mucositis for modified dose level four.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Sullivan, M.D., Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/